CLINICAL TRIAL: NCT07213895
Title: Randomized, Single Oral Dose, Two-period, Two Sequence, Open-label, Crossover, Bioequivalence Study to Compare Empagliflozin-Linagliptin-Metformin XR Tablet 25mg/ 5mg/1000mg (25mg Empagliflozin /5mg Linagliptin /1000mg Metformin Hydrochloride) Versus Trijardy® XR Tablets (25mg Empagliflozin /5mg Linagliptin /1000mg Metformin Hydrochloride), in Healthy Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study to Compare Empagliflozin/Linagliptin/Metformin HCL 25mg/5mg/1000mg Extended-Release Tablets Versus Trijardy® XR Extended Release Film Coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1392-2025, V.01
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin/Linagliptin/Metformin HCL Extended Release Tablets (Experimental): Empagliflozin/Linagliptin/Metformin HCL 25mg/5mg/1000mg Extended Release Tablets
  Interventions: Drug: Empagliflozin/Linagliptin/Metformin HCL; Drug: Trijardy® XR Extended release film coated tablets
- Trijardy® XR Extended release film coated tablets (Active Comparator): Trijardy® 25mg/5mg/1000mg Extended release film coated tablets
  Interventions: Drug: Empagliflozin/Linagliptin/Metformin HCL; Drug: Trijardy® XR Extended release film coated tablets

INTERVENTIONS:
Drug: Empagliflozin/Linagliptin/Metformin HCL — One Empagliflozin/Linagliptin/Metformin HCL 25mg/5mg/1000mg extended release film-coated tablet
Drug: Trijardy® XR Extended release film coated tablets — One Trijardy® 25mg/5mg/1000mg Extended Release Tablets

SUMMARY:
Randomized, Single Oral Dose, Two-period, Two Sequence, Open-label, Crossover, Bioequivalence Study to Compare Empagliflozin-Linagliptin-Metformin XR Tablet 25mg/ 5mg/1000mg (25mg Empagliflozin /5mg Linagliptin /1000mgMetformin Hydrochloride) Versus Trijardy® XR Tablets (25mg Empagliflozin /5mg Linagliptin /1000mg Metformin Hydrochloride), in Healthy Subjects Under Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is caucasian & aged between eighteen & fifty years (18-50), both inclusive.
* The subject is within the limits for his/her height & weight as defined by the body mass index range (18.5 - 30.0 kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative serum pregnancy test and the woman is using two reliable contraception methods and should be non-lactating.
* The subject has normal cardiovascular system & normal ECG with normal QT interval corrected for heart rate according to Bazett's formula.
* The subject's kidney and liver (AST & ALT enzymes) function tests are within normal range. (Creatinine is accepted if below the reference range after being evaluated by the clinical investigator as clinically not significant).
* The subject's HbA1c test result is within normal range (HbA1c is accepted if below the reference range after being evaluated by the clinical investigator as clinically not significant.)
* The subject's fasting blood glucose level is ≥ 70 mg/dL before dosing.
* The subject Hematology test results are within normal range & RBC indices are within 5% of the normal range.

Exclusion Criteria:

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is on special diet (for example subject is vegetarian).
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing in both study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit/ orange containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* The subject has consumed drugs that may affect pharmacological/ pharmacokinetic properties of Empagliflozin/Linagliptin/Metformin hydrochloride (for example: Ethanol, Ioversol, Probenecid, Iodinated contrast media, Rifampicin, Gemfibrozil, Glimepiride, Sitagliptin, Warfarin, Verapamil, Ramipril, Torasemide, Hydrochlorothiazide, Lithium, Cimetidine, apalutamide, Benazepril, Idelalisib, Ivosidenib, Lasmiditan, Methylene blue, Ranolazine, Selegiline, Tafenoquine, Tedizolid, Tranylcypromine, Tucatinib, Voxelotor, Sulphonylureas, Ritonavir, Dolutegravir, Cimetidine, Trimethoprime, Isavuconazonium, Crizotinib, Olaparib, Trimethoprime, Vandetanib, Isavuconazole, Glucocorticoids, Insulin and insulin secretagogues (Sulphonylureas)) two weeks before and after the study and during the study.
* The subject has a history of ketone in urine, presence of any type of acute metabolic acidosis (such as lactic acidosis).

Note: Subjects, who were screened for another study and were not enrolled, might be recruited for this study provided they meet the acceptance criteria of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
For Empagliflozin & Linagliptin & Metformin; Maximum concentration obtained (Cmax) | 72 hours
  two-sides 90% CI for the test to reference ratio of the population means is within 80.00-125.00% for each of the Ln-transformed data Cmax
For Linagliptin; AUC from time 0 to last collection time (AUC0 - 72 due to Linagliptin long half-life) | 72 hours
  two-sides 90% CI for the test to reference ratio of the population means is within 80.00-125.00% for each of the Ln-transformed data AUC
For Metformin; AUC from time 0 to last collection time (AUC0-t) | 72 hours
  two-sides 90% CI for the test to reference ratio of the population means is within 80.00-125.00% for each of the Ln-transformed data AUC

SECONDARY OUTCOMES:
For Empagliflozin & Linagliptin & Metformin; Time to reach maximum concentration Cmax (Tmax) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- ACDIMA Center, Amman, Jordan